CLINICAL TRIAL: NCT06811571
Title: A Study of the Effectiveness of a Mobile-based Early Intervention on Adolescent Hazardous Gaming
Brief Title: A Study of the Effectiveness of an Early Intervention on Adolescent Hazardous Gaming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NZhong-007
Record Dates: First submitted 2024-07-16; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-06

CONDITIONS: Gaming Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the intervention group (Experimental): The mobile-based early intervention on adolescent hazardous gaming was implemented through WeChat, a popular multipurpose social-networking app in China. The mini-program regularly delivered contents to the users' WeChat homepage, reminding them to timely complete the interventions. The completion status of the users was collected and sent to the backend intervention provider. The intervention group received the one-month intervention.
  Interventions: Behavioral: the mobile-based early intervention
- the control group (No Intervention): The control group did not receive the intervention. Both two groups accepted the assessments at baseline and two months after the intervention.

INTERVENTIONS:
Behavioral: the mobile-based early intervention — The theoretical framework of the intervention was based on Cognitive Behavior Therapy (CBT). We designed three modules, which were the Gaming behavior management, the Gaming cognition establishment and the Early intervention on risk and protective factors. The interventions included self-monitoring questionnaires, scientific popular articles, and online lectures.
  Arms: the intervention group

SUMMARY:
The investigators established a mobile-based early intervention on adolescent hazardous gaming and verified its effectiveness.

DETAILED DESCRIPTION:
Hazardous gaming is the precursor of gaming disorder. Early intervention on hazardous gaming is an effective strategy to prevent gaming disorder. Currently, there are few evidence-based early interventions, particularly the technology-based approaches with the advantage of user-friendliness. This study developed a mobile-based early intervention program based on cognitive-behavioral therapy (CBT) for adolescent hazardous gaming. In order to verify the effectiveness of the intervention, adolescent participants were recruited and divided into two groups. The intervention group received the one-month intervention, while the control group did not. Both groups accepted the assessments at baseline and two months after the intervention. Comparative analysis was carried out between the two groups and two time points, primarily on the severity of gaming disorder, gaming hours, gaming frequency, anxiety, depression and self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of hazardous gaming defined in the ICD-11 (2) Fully comprehending the research's purpose and procedures and signing the informed consent

Exclusion Criteria:

* (1)Serious physical illness or intellectual disability (2) Clinical diagnosis of gaming disorder (3) Not completing all the interventions or assessments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the severity of gaming disorder | baseline, two months after intervention
  Measured by Gaming Disorder Screening Scale

SECONDARY OUTCOMES:
average daily gaming hours | baseline, two months after intervention
  self-reported average hours spent gaming per day
frequency of gaming sessions | baseline, two months after intervention
  self-reported number of gaming sessions per week
anxiety severity | baseline, two months after intervention
  Measured by: Generalized Anxiety Disorder 7-item (GAD-7) Scale Scale Range: 0 to 21 (higher scores indicate worse anxiety)
depression severity | baseline, two months after intervention
  Measured by: Patient Health Questionnaire-9 (PHQ-9) Scale Range: 0 to 27 (higher scores indicate worse depression)
self-esteem | baseline, two months after intervention
  Measured by: Rosenberg Self-Esteem Scale (SES) Scale Range: 0 to 30 (higher scores indicate better self-esteem)

CONTACTS AND LOCATIONS:
Overall Officials: Na Zhong, MD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China